CLINICAL TRIAL: NCT04068688
Title: Tailoring Treatment Targets for Early Autism Intervention in Africa
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: University of Cape Town (Other); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: Pro00103045; 1R21MH120696 (NIH)
Record Dates: First submitted 2019-08-20; First posted 2019-08-28 (Actual); Results first posted 2022-12-02 (Actual); Last update posted 2022-12-02 (Actual); Status verified 2022-11

CONDITIONS: Autism Spectrum Disorder
Keywords: NDBI; Autism
MeSH Terms: conditions — Autism Spectrum Disorder; Autistic Disorder

STUDY DESIGN:
Intervention Model Description: Note the autism group will be the only group to receive intervention. The typically developing and developmental delay group will receive one baseline assessment, and no intervention. COVID-19 necessitated a pivot from in-person to telehealth coaching.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Caregiver-Child Dyads with ASD (Autism Spectrum Disorder) (Experimental): Participants in this arm will be caregivers of and children with ASD.
  Interventions: Behavioral: Early Start Denver Model (ESDM)
- Children with typical development (No Intervention): Participants in this arm will be children with typical development.
- Children with developmental delay (No Intervention): Participants in this arm will be children with developmental delay.
- Caregiver-Child Dyads with ASD (Autism Spectrum Disorder) Telehealth Adaptation (Experimental): Participants in this arm will be caregivers of and children with ASD receiving telehealth intervention (adaptation due to COVID-19 restrictions).
  Interventions: Behavioral: Telehealth coaching
- Early Childhood Development (ECD) Practitioners and ECD Practitioner School Supervisors (No Intervention): The ECD worker and/or school supervisor are 1) employed by our participating recruitment partners (Western Cape Education Department Schools) and 2) involved in delivery of the caregiver coaching sessions, either in person or remotely.
- Early Start Denver Model (ESDM) Supervisors (No Intervention): The local supervisors are 1) trained ESDM therapist, 2) supervise weekly coaching sessions in the schools, and/or 3) supervise remote intervention delivery sessions.

INTERVENTIONS:
Behavioral: Early Start Denver Model (ESDM) — Twelve one hour sessions, skill is introduced by "Help is in your hands" Community ESDM videos. Session skills include specific strategies caregivers can use to increase their child's attention to people and their child's communication; strategies to identify, create and use joint activity routines to engage with and teach their child; in addition to ways to use the ABCs of learning to teach their child new behaviors. "Help is in your hands" Community ESDM materials also provide video examples of other caregivers using the session skill with their child. The early childhood development practitioner then coaches the caregiver in the session skill, in at least two activities. The goal of coaching was to provide enough support for the caregiver to experience success in implementing the new skill with their child. Coaching is followed by caregiver reflection and a discussion of generalization of the new skill across various daily activities, using a daily activities visual aid.
  Arms: Caregiver-Child Dyads with ASD (Autism Spectrum Disorder)
Behavioral: Telehealth coaching — The telehealth coaching intervention was informed by the Community-Early Start Denver Model (C-ESDM) materials. Twelve session-specific visuals with simple-text (for caregivers) and session scripts (for non-specialist coaches) were developed by the research team. Over 12, 1-hour asynchronous caregiver coaching sessions that are delivered by non-specialists, caregivers were coached in strategies to increase child attention to their social world, increase child communication, create and build joint activity routines, and understand and use the ABCs to support the development of new behaviors. The session itself being delivered via phone. Prior to the coaching session staff shared session materials with the family via WhatsApp. Prior to the session the caregiver shared a 6-min video of an interaction with their child. During the session, the caregiver and coach reviewed the video, and the caregiver completed a self-reflection checklist.
  Arms: Caregiver-Child Dyads with ASD (Autism Spectrum Disorder) Telehealth Adaptation

SUMMARY:
Naturalistic Developmental Behavioral Interventions (NDBIs), an evidence-based early autism spectrum disorder (ASD) intervention approach, target key behaviors that help language development. While efforts to use NDBIs are increasing worldwide, important gaps in our knowledge remain on whether the behaviors targeted by NDBIs are cross-culturally valid. This study in South Africa, a multi-cultural setting, will provide critical information on NDBI treatment targets and a novel digital outcome measure of treatment response.

COVID-19 adaptations: We aim to develop and implement telehealth NDBI coaching and utilize a mixed methods approach to gather implementation and preliminary effectiveness data on the telehealth intervention.

DETAILED DESCRIPTION:
COVID-19 has significantly impacted autism spectrum disorder (ASD) clinical research and disrupted access to intervention services for children and families globally. In this ongoing study in Cape Town South Africa, a caregiver coaching Naturalistic Developmental Behavioral Intervention (NDBI) for young children with ASD has been adapted for implementation by non-specialists and implementation and clinical outcomes are being evaluated. For ongoing clinical trials, the University of Cape Town Institutional Review Board (IRB) has encouraged researchers to switch to a virtual platform, where possible. Telehealth caregiver coaching is cost-effective, increases access to rural and underserved populations, and improves understanding of family home and caregiving routines. We aim to develop and implement telehealth NDBI coaching and utilize a mixed methods approach and a longitudinal pre-post design to gather implementation and preliminary effectiveness data on the telehealth intervention.

ELIGIBILITY:
Inclusion Criteria:

1. For ASD, DD, TD groups

   * Subject family speaks isiXhosa, Afrikaans, or English
   * Child's ethnicity/race is African or Coloured (A South African term for individuals with mixed racial heritage)
   * Child lives within an area served by the recruitment sites
2. For the ASD group only:

   * Child meets criteria for an ASD diagnosis based upon DSM-5 (Diagnostic and Statistical Manual of Mental Disorders) criteria and informed by the ADOS-2 (Autism Diagnostic Observation Schedule) administered by research reliable raters
   * Caregiver is at least 18 years old
3. For the developmental delay (DD) group only:

   * Child screens positive on the Ten Questions and negative for ASD on the ABC
   * Child has been diagnosed with developmental delay by a developmental pediatrician
4. For the typically developing (TD) group only:

   -Child screens negative on the Ten Questions and negative for ASD on the ABC
5. For the Early Childhood Development (ECD) Practitioners and Early Childhood Development Practitioner School Supervisors group:

   * Employed by participating recruitment partners (Western Cape Education Department Schools)
   * Involved in delivery of the caregiver coaching sessions, either in person or remotely
6. For the Early Start Denver Model (ESDM) supervisors group:

   * Trained ESDM therapist
   * Supervise weekly coaching sessions in the schools, and/or
   * Supervise remote intervention delivery sessions

Exclusion Criteria:

1. For all groups (ASD, DD, TD)

   * Significant sensory or motor impairment
   * Major physical abnormalities
   * History of serious head injury and/or neurological disease
2. For the ASD group:

   * Presence of a neurological disorder of known etiology (for e.g., Downs Syndrome)
   * Caregiver-child dyad unable to attend assessments and 12 coaching sessions
3. For the developmental delay (DD) group

   -Autism diagnosis based on DSM 5 criteria
4. For typically developing (TD group:

   * Autism diagnosis based on DSM 5 criteria

Ages: 18 Months to 72 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 73 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2021-08-26 (Actual); Study Completion 2021-08-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lauren Franz, MB, CHB, Principal Investigator — Duke University
Locations (1):
- University of Cape Town, Cape Town, West Cape, South Africa

IPD SHARING:
Plan to Share IPD: Yes
All individual-level descriptive data will be submitted to the NIH/NIMH (National Institute of Mental Health) data repositories on a quarterly. Submission of all other experimental data will occur after the primary objectives of the R21 have been met. Prior to submission, dedicated research staff will review accuracy and conduct additional manual and automated checks for presence of protected health information (PHI) in the submitted data. Submissions will include protocols, questionnaires, study manuals, variables measured, and any other necessary documentation. All submitted data (both descriptive/raw and analyzed data) will be made available for access by members of the research community according to the provisions defined in the NDAR (National Database for Autism Research) and the NIH/NIMH Data Repositories Data Sharing Policy. All research data will be made accessible to other researchers within four months of submission, allowing sufficient time to complete QA/QC procedures.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: As per NDAR requirements

RESULTS

PARTICIPANT FLOW:
Recruitment Details: ASD caregiver-child dyads were recruited from Western Cape Department of Education Autism Schools; children with developmental delay from Neurodevelopmental Clinics at Red Cross Children's Hospital; typically developing children from ECD Centers. ASD caregiver-child dyads could opt to continue with Telehealth intervention when COVID restrictions were implemented. Participants recruited March 2020-March 2021 received telehealth intervention.
Pre-assignment Details: One participant from the Children with Typical Development group was deemed ineligible post-enrollment.
Groups:
- Caregiver-Child Dyads With ASD (In-person Intervention ONLY) - Caregivers: Participants in this arm will be caregivers of children with ASD. Early Start Denver Model (ESDM): Twelve one hour sessions, skill is introduced by "Help is in your hands" Community ESDM videos. Session skills include specific strategies caregivers can use to increase their child's attention to people and their child's communication; strategies to identify, create and use joint activity routines to engage with and teach their child; in addition to ways to use the ABCs of learning to teach their child new behaviors. "Help is in your hands" Community ESDM materials also provide video examples of other caregivers using the session skill with their child. The early childhood development practitioner then coaches the caregiver in the session skill, in at least two activities. The goal of coaching was to provide enough support for the caregiver to experience success in implementing the new skill with their child. Coaching is followed by caregiver reflection and a discussion of generalization of the new skill across various daily activities, using a daily activities visual aid.
- Caregiver-Child Dyads With ASD (In-person Intervention ONLY) - Children: Participants in this arm will be children with ASD. Early Start Denver Model (ESDM): Twelve one hour sessions, skill is introduced by "Help is in your hands" Community ESDM videos. Session skills include specific strategies caregivers can use to increase their child's attention to people and their child's communication; strategies to identify, create and use joint activity routines to engage with and teach their child; in addition to ways to use the ABCs of learning to teach their child new behaviors. "Help is in your hands" Community ESDM materials also provide video examples of other caregivers using the session skill with their child. The early childhood development practitioner then coaches the caregiver in the session skill, in at least two activities. The goal of coaching was to provide enough support for the caregiver to experience success in implementing the new skill with their child. Coaching is followed by caregiver reflection and a discussion of generalization of the new skill across various daily activities, using a daily activities visual aid.
- Caregiver-Child Dyads With ASD (In-person, Then Telehealth Intervention) - Caregivers: Participants in this arm will be caregivers of children with ASD who began the intervention in-person and moved to telehealth due to COVID-19 restrictions.
  In-person: Twelve 1-hour sessions, skill is introduced by "Help is in your hands" Community Early Start Denver Model (C-ESDM) videos. Skills include specific strategies caregivers can use to increase their child's attention to people and their child's communication; strategies to identify, create and use joint activity routines to engage with and teach their child; in addition to ways to use the ABCs of learning to teach their child new behaviors. The ECD practitioner then coaches the caregiver in at least two activities. Coaching is followed by caregiver reflection and a discussion of generalization of the new skill using a daily activities visual aid.
  Telehealth coaching: The telehealth coaching intervention was informed by the C-ESDM materials. Twelve session-specific visuals with simple-text (for caregivers) and session scripts (for non-specialist coaches) were developed by the research team. Over 12, 1-hour asynchronous caregiver coaching sessions that are delivered by non-specialists, caregivers were coached as above (via phone). Prior to the coaching session staff shared session materials with the family via WhatsApp and the caregiver shared a 6-min video of an interaction with their child. During the session, the caregiver and coach reviewed the video, and the caregiver completed a self-reflection checklist.
- Caregiver-Child Dyads With ASD (In-person, Then Telehealth Intervention) - Children: Participants in this arm will be children with ASD who began the intervention in-person and moved to telehealth due to COVID-19 restrictions.
  In-person: Twelve 1-hour sessions, skill is introduced by "Help is in your hands" Community Early Start Denver Model (C-ESDM) videos. Skills include specific strategies caregivers can use to increase their child's attention to people and their child's communication; strategies to identify, create and use joint activity routines to engage with and teach their child; in addition to ways to use the ABCs of learning to teach their child new behaviors. The ECD practitioner then coaches the caregiver in at least two activities. Coaching is followed by caregiver reflection and a discussion of generalization of the new skill using a daily activities visual aid.
  Telehealth coaching: The telehealth coaching intervention was informed by the C-ESDM materials. Twelve session-specific visuals with simple-text (for caregivers) and session scripts (for non-specialist coaches) were developed by the research team. Over 12, 1-hour asynchronous caregiver coaching sessions that are delivered by non-specialists, caregivers were coached as above (via phone). Prior to the coaching session staff shared session materials with the family via WhatsApp and the caregiver shared a 6-min video of an interaction with their child. During the session, the caregiver and coach reviewed the video, and the caregiver completed a self-reflection checklist.
- Caregiver-Child Dyads With ASD (Telehealth Intervention ONLY) - Caregivers: Participants in this arm will be caregivers of children with ASD receiving telehealth intervention (adaptation due to COVID-19 restrictions).
  Telehealth coaching: The telehealth coaching intervention was informed by the Community-Early Start Denver Model (C-ESDM) materials. Twelve session-specific visuals with simple-text (for caregivers) and session scripts (for non-specialist coaches) were developed by the research team. Over 12, 1-hour asynchronous caregiver coaching sessions that are delivered by non-specialists, caregivers were coached in strategies to increase child attention to their social world, increase child communication, create and build joint activity routines, and understand and use the ABCs to support the development of new behaviors. The session itself being delivered via phone. Prior to the coaching session staff shared session materials with the family via WhatsApp. Prior to the session the caregiver shared a 6-min video of an interaction with their child. During the session, the caregiver and coach reviewed the video, and the caregiver completed a self-reflection checklist.
- Caregiver-Child Dyads With ASD (Telehealth Intervention ONLY) - Children: Participants in this arm will be children with ASD receiving telehealth intervention (adaptation due to COVID-19 restrictions).
  Telehealth coaching: The telehealth coaching intervention was informed by the Community-Early Start Denver Model (C-ESDM) materials. Twelve session-specific visuals with simple-text (for caregivers) and session scripts (for non-specialist coaches) were developed by the research team. Over 12, 1-hour asynchronous caregiver coaching sessions that are delivered by non-specialists, caregivers were coached in strategies to increase child attention to their social world, increase child communication, create and build joint activity routines, and understand and use the ABCs to support the development of new behaviors. The session itself being delivered via phone. Prior to the coaching session staff shared session materials with the family via WhatsApp. Prior to the session the caregiver shared a 6-min video of an interaction with their child. During the session, the caregiver and coach reviewed the video, and the caregiver completed a self-reflection checklist.
- Children With Typical Development: Participants in this arm will be children with typical development. No intervention.
- Children With Developmental Delay: Participants in this arm will be children with developmental delay. No intervention.
Period: Overall Study
Arm/Group | Caregiver-Child Dyads With ASD (In-person Intervention ONLY) - Caregivers | Caregiver-Child Dyads With ASD (In-person Intervention ONLY) - Children | Caregiver-Child Dyads With ASD (In-person, Then Telehealth Intervention) - Caregivers | Caregiver-Child Dyads With ASD (In-person, Then Telehealth Intervention) - Children | Caregiver-Child Dyads With ASD (Telehealth Intervention ONLY) - Caregivers | Caregiver-Child Dyads With ASD (Telehealth Intervention ONLY) - Children | Children With Typical Development | Children With Developmental Delay | Early Childhood Development (ECD) Practitioners and ECD Practitioner School Supervisors | Early Start Denver Model (ESDM) Supervisors
Started | 17 | 17 | 2 | 2 | 12 | 12 | 2 | 1 | 4 | 3
Completed | 8 | 8 | 2 | 2 | 7 | 7 | 2 | 1 | 3 | 3
Not Completed | 9 | 9 | 0 | 0 | 5 | 5 | 0 | 0 | 1 | 0
Not completed — Lost to Follow-up | 1 | 1 | 0 | 0 | 5 | 5 | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Unable to complete intervention due to COVID-19 restrictions | 7 | 7 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Caregiver-Child Dyads With ASD (In-person Intervention ONLY) - Caregivers | Caregiver-Child Dyads With ASD (In-person Intervention ONLY) - Children | Caregiver-Child Dyads With ASD (In-person, Then Telehealth Intervention) - Caregivers | Caregiver-Child Dyads With ASD (In-person, Then Telehealth Intervention) - Children | Caregiver-Child Dyads With ASD (Telehealth Intervention ONLY) - Caregivers | Caregiver-Child Dyads With ASD (Telehealth Intervention ONLY) - Children | Children With Typical Development | Children With Developmental Delay | Early Childhood Development (ECD) Practitioners and ECD Practitioner School Supervisors | Early Start Denver Model (ESDM) Supervisors | Total
Number analyzed (Participants) | 17 | 17 | 2 | 2 | 12 | 12 | 2 | 1 | 4 | 3 | 72
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Caregivers only. Data not collected on ECD Practitioners and ECD Practitioner School Supervisors or ESDM Supervisors groups.
  years
    number analyzed (Participants) | 17 | 0 | 2 | 0 | 12 | 0 | 0 | 0 | 0 | 0 | 31
    (all) | 36.12 (9.60) |  | 36 (7.07) |  | 35.5 (7.52) |  |  |  |  |  | 35.92 (8.56)
Age, Continuous [Mean (Standard Deviation); unit: months] — Population: Children only. Data not collected on ECD Practitioners and ECD Practitioner School Supervisors or ESDM Supervisors groups.
  months
    number analyzed (Participants) | 0 | 17 | 0 | 2 | 0 | 12 | 2 | 1 | 0 | 0 | 34
    (all) |  | 50.19 (9.66) |  | 40.5 (17.68) |  | 51.25 (16.94) | 41 (7.07) | 18 (0) |  |  | 48.07 (13.42)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 3 | 1 | 1 | 10 | 2 | 1 | 1 | 4 | 3 | 37
  Male | 6 | 14 | 1 | 1 | 2 | 10 | 1 | 0 | 0 | 0 | 35
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 17 | 17 | 2 | 2 | 12 | 12 | 2 | 1 | 4 | 3 | 72
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 4 | 5 | 2 | 2 | 0 | 0 | 1 | 1 | 0 | 1 | 16
  White | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2
  More than one race | 9 | 10 | 0 | 0 | 7 | 7 | 1 | 0 | 3 | 0 | 37
  Unknown or Not Reported | 3 | 2 | 0 | 0 | 4 | 4 | 0 | 0 | 1 | 0 | 14
Region of Enrollment [Count of Participants; unit: Participants]
  South Africa | 17 | 17 | 2 | 2 | 12 | 12 | 2 | 1 | 4 | 3 | 72

OUTCOME MEASURES:

1. Primary Outcome: Supported Joint Engagement Measured by the Joint Engagement Rating Inventory (JERI)
Description: Child engagement states measured by the Joint Engagement Rating Inventory (JERI) ; in the ASD group; the typically developing group; and the developmental delay group. Joint Engagement Rating Inventory contains eighteen 7-point Likert scale items that characterized various aspects of joint engagement. The items were designed to span the range of possibilities likely to be observed during interactions with 18- to 30-month-old TD children as well as similarly aged and older children with developmental difficulties, including ASD. A rating of 1 indicates a very low rating and no time spent in that engagement state, 4 is the midpoint indicating the moderate time and quality of episodes in an engagement state, and 7 indicates a very high rating and high-quality engagement.
Time Frame: Baseline and Follow-up (after 12 intervention sessions, up to 3 months)
Population: Participants who completed the study. Only applicable to Caregiver-Child Dyads With ASD, Children with typical development, and Children with developmental delay groups. Data only collected at baseline for Children with Typical Development and Children with Developmental Delay.
Measure: Median (Full Range); unit: score on a scale
Groups:
- Caregiver-Child Dyads With ASD (In-person Intervention ONLY): Participants in this arm will be caregivers of and children with ASD. Early Start Denver Model (ESDM): Twelve one hour sessions, skill is introduced by "Help is in your hands" Community ESDM videos. Session skills include specific strategies caregivers can use to increase their child's attention to people and their child's communication; strategies to identify, create and use joint activity routines to engage with and teach their child; in addition to ways to use the ABCs of learning to teach their child new behaviors. "Help is in your hands" Community ESDM materials also provide video examples of other caregivers using the session skill with their child. The early childhood development practitioner then coaches the caregiver in the session skill, in at least two activities. The goal of coaching was to provide enough support for the caregiver to experience success in implementing the new skill with their child. Coaching is followed by caregiver reflection and a discussion of generalization of the new skill across various daily activities, using a daily activities visual aid.
- Caregiver-Child Dyads With ASD (Telehealth Intervention): Participants in this arm will be caregivers of and children with ASD receiving only telehealth intervention (adaptation due to COVID-19 restrictions) or as a continuation of in-person intervention.
  Telehealth coaching: The telehealth coaching intervention was informed by the Community-Early Start Denver Model (C-ESDM) materials. Twelve session-specific visuals with simple-text (for caregivers) and session scripts (for non-specialist coaches) were developed by the research team. Over 12, 1-hour asynchronous caregiver coaching sessions that are delivered by non-specialists, caregivers were coached in strategies to increase child attention to their social world, increase child communication, create and build joint activity routines, and understand and use the ABCs to support the development of new behaviors. The session itself being delivered via phone. Prior to the coaching session staff shared session materials with the family via WhatsApp. Prior to the session the caregiver shared a 6-min video of an interaction with their child. During the session, the caregiver and coach reviewed the video, and the caregiver completed a self-reflection checklist.
Arm/Group | Caregiver-Child Dyads With ASD (In-person Intervention ONLY) | Caregiver-Child Dyads With ASD (Telehealth Intervention) | Children With Typical Development | Children With Developmental Delay
Number analyzed (Participants) | 8 | 9 | 2 | 1
score on a scale
  Baseline | 6 [3 to 6] | 4 [3 to 6] | 2 [2 to 2] | 4 [4 to 4]
  Follow-up: number analyzed (Participants) | 8 | 9 | 0 | 0
  Follow-up | 5.5 [4 to 6] | 5 [1 to 6] |  |
Statistical Analysis 1: Comparison: Caregiver-Child Dyads With ASD (In-person Intervention ONLY); Test type: Other; p = 1.00, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Caregiver-Child Dyads With ASD (Telehealth Intervention); Test type: Other; p = 0.914, Wilcoxon (Mann-Whitney)

2. Primary Outcome: Coordinated Joint Engagement Measured by the Joint Engagement Rating Inventory (JERI)
Description: Child engagement states measured by the Joint Engagement Rating Inventory (JERI) in the ASD group; the typically developing group; and the developmental delay group. Joint Engagement Rating Inventory contains eighteen 7-point Likert scale items that characterized various aspects of joint engagement. The items were designed to span the range of possibilities likely to be observed during interactions with 18- to 30-month-old TD children as well as similarly aged and older children with developmental difficulties, including ASD. A rating of 1 indicates a very low rating and no time spent in that engagement state, 4 is the midpoint indicating the moderate time and quality of episodes in an engagement state, and 7 indicates a very high rating and high-quality engagement.
Time Frame: Baseline and Follow-up (after 12 intervention sessions, up to 3 months)
Population: as for outcome 1
Measure: Median (Full Range); unit: score on a scale
Groups:
- Caregiver-Child Dyads With ASD (Telehealth Intervention): Participants in this arm will be caregivers of and children with ASD receiving telehealth intervention (adaptation due to COVID-19 restrictions) or as a continuation of in-person intervention.
  Telehealth coaching: The telehealth coaching intervention was informed by the Community-Early Start Denver Model (C-ESDM) materials. Twelve session-specific visuals with simple-text (for caregivers) and session scripts (for non-specialist coaches) were developed by the research team. Over 12, 1-hour asynchronous caregiver coaching sessions that are delivered by non-specialists, caregivers were coached in strategies to increase child attention to their social world, increase child communication, create and build joint activity routines, and understand and use the ABCs to support the development of new behaviors. The session itself being delivered via phone. Prior to the coaching session staff shared session materials with the family via WhatsApp. Prior to the session the caregiver shared a 6-min video of an interaction with their child. During the session, the caregiver and coach reviewed the video, and the caregiver completed a self-reflection checklist.
Arm/Group | Caregiver-Child Dyads With ASD (In-person Intervention ONLY) | Caregiver-Child Dyads With ASD (Telehealth Intervention) | Children With Typical Development | Children With Developmental Delay
Number analyzed (Participants) | 8 | 9 | 2 | 1
score on a scale
  Baseline | 1 [1 to 3] | 1 [1 to 2] | 6 [6 to 6] | 2 [2 to 2]
  Follow-up: number analyzed (Participants) | 8 | 9 | 0 | 0
  Follow-up | 1 [1 to 4] | 1 [1 to 3] |  |
Statistical Analysis 1: Comparison: Caregiver-Child Dyads With ASD (In-person Intervention ONLY); Test type: Other; p = 0.655, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Caregiver-Child Dyads With ASD (Telehealth Intervention); Test type: Other; p = 0.564, Wilcoxon (Mann-Whitney)

3. Primary Outcome: Symbol-infused Joint Engagement Measured by the Joint Engagement Rating Inventory (JERI)
Description: as for outcome 2
Time Frame: Baseline and Follow-up (after 12 intervention sessions, up to 3 months)
Population: as for outcome 1
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Caregiver-Child Dyads With ASD (In-person Intervention ONLY) | Caregiver-Child Dyads With ASD (Telehealth Intervention) | Children With Typical Development | Children With Developmental Delay
Number analyzed (Participants) | 8 | 9 | 2 | 1
score on a scale
  Baseline | 2 [1 to 3] | 2 [1 to 4] | 6.5 [6 to 7] | 2 [2 to 2]
  Follow-up: number analyzed (Participants) | 8 | 9 | 0 | 0
  Follow-up | 3 [1 to 4] | 1 [1 to 5] |  |
Statistical Analysis 1: Comparison: Caregiver-Child Dyads With ASD (In-person Intervention ONLY); Test type: Other; p = 0.014, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Caregiver-Child Dyads With ASD (Telehealth Intervention); Test type: Other; p = 0.705, Wilcoxon (Mann-Whitney)

4. Primary Outcome: Fluency and Connectedness Measured by the Joint Engagement Rating Inventory (JERI)
Description: Caregiver-child dyadic exchanges measured by the Joint Engagement Rating Inventory (JERI) in the ASD group. Joint Engagement Rating Inventory contains eighteen 7-point Likert scale items that characterized various aspects of joint engagement. The items were designed to span the range of possibilities likely to be observed during interactions with 18- to 30-month-old TD children as well as similarly aged and older children with developmental difficulties, including ASD. A rating of 1 indicates no interaction between the dyad, a rating of 7 indicates a balanced dyadic exchange that flows naturally back and forth.
Time Frame: Baseline and Follow-up (after 12 intervention sessions, up to 3 months)
Population: as for outcome 1
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Caregiver-Child Dyads With ASD (In-person Intervention ONLY) | Caregiver-Child Dyads With ASD (Telehealth Intervention) | Children With Typical Development | Children With Developmental Delay
Number analyzed (Participants) | 8 | 9 | 2 | 1
score on a scale
  Baseline | 4 [3 to 5] | 4 [3 to 6] | 6 [6 to 6] | 3 [3 to 3]
  Follow-up: number analyzed (Participants) | 8 | 9 | 0 | 0
  Follow-up | 5 [3 to 6] | 5 [2 to 6] |  |
Statistical Analysis 1: Comparison: Caregiver-Child Dyads With ASD (In-person Intervention ONLY); Test type: Other; p = 0.096, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Caregiver-Child Dyads With ASD (Telehealth Intervention); Test type: Other; p = 0.732, Wilcoxon (Mann-Whitney)

5. Primary Outcome: Shared Routines and Rituals Measured by the Joint Engagement Rating Inventory (JERI)
Description: as for outcome 4
Time Frame: Baseline and Follow-up (after 12 intervention sessions, up to 3 months)
Population: as for outcome 1
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Caregiver-Child Dyads With ASD (In-person Intervention ONLY) | Caregiver-Child Dyads With ASD (Telehealth Intervention) | Children With Typical Development | Children With Developmental Delay
Number analyzed (Participants) | 8 | 9 | 2 | 1
score on a scale
  Baseline | 1 [1 to 2] | 1 [1 to 5] | 1 [1 to 1] | 1 [1 to 1]
  Follow-up: number analyzed (Participants) | 8 | 9 | 0 | 0
  Follow-up | 1 [1 to 3] | 1 [1 to 3] |  |
Statistical Analysis 1: Comparison: Caregiver-Child Dyads With ASD (In-person Intervention ONLY); Test type: Other; p = 1.00, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Caregiver-Child Dyads With ASD (Telehealth Intervention); Test type: Other; p = 0.705, Wilcoxon (Mann-Whitney)

6. Primary Outcome: Scaffolding Measured by the Joint Engagement Rating Inventory (JERI)
Description: Caregiver strategies measured by the Joint Engagement Rating Inventory (JERI) in the ASD group. Joint Engagement Rating Inventory contains eighteen 7-point Likert scale items that characterized various aspects of joint engagement. The items were designed to span the range of possibilities likely to be observed during interactions with 18- to 30-month-old TD children as well as similarly aged and older children with developmental difficulties, including ASD. A rating of 1 indicates that the caregiver rarely uses the caregiver strategy to support the child's activity and language. A rating of 7 indicates that the caregiver frequently uses appropriate strategies to support and expand their child's activity and language.
Time Frame: Baseline and Follow-up (after 12 intervention sessions, up to 3 months)
Population: as for outcome 1
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Caregiver-Child Dyads With ASD (In-person Intervention ONLY) | Caregiver-Child Dyads With ASD (Telehealth Intervention) | Children With Typical Development | Children With Developmental Delay
Number analyzed (Participants) | 8 | 9 | 2 | 1
score on a scale
  Baseline | 5 [3 to 6] | 4 [3 to 5] | 5 [4 to 6] | 2 [2 to 2]
  Follow-up: number analyzed (Participants) | 8 | 9 | 0 | 0
  Follow-up | 5 [3 to 7] | 4 [3 to 6] |  |
Statistical Analysis 1: Comparison: Caregiver-Child Dyads With ASD (In-person Intervention ONLY); Test type: Other; p = 0.442, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Caregiver-Child Dyads With ASD (Telehealth Intervention); Test type: Other; p = 0.458, Wilcoxon (Mann-Whitney)

7. Primary Outcome: Following in on a Child's Focus Measured by the Joint Engagement Rating Inventory (JERI)
Description: as for outcome 6
Time Frame: Baseline and Follow-up (after 12 intervention sessions, up to 3 months)
Population: as for outcome 1
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Caregiver-Child Dyads With ASD (In-person Intervention ONLY) | Caregiver-Child Dyads With ASD (Telehealth Intervention) | Children With Typical Development | Children With Developmental Delay
Number analyzed (Participants) | 8 | 9 | 2 | 1
score on a scale
  Baseline | 5 [3 to 7] | 5 [3 to 7] | 5 [4 to 6] | 2 [2 to 2]
  Follow-up: number analyzed (Participants) | 8 | 9 | 0 | 0
  Follow-up | 6 [3 to 7] | 5 [3 to 6] |  |
Statistical Analysis 1: Comparison: Caregiver-Child Dyads With ASD (In-person Intervention ONLY); Test type: Other; p = 0.35, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Caregiver-Child Dyads With ASD (Telehealth Intervention); Test type: Other; p = 0.68, Wilcoxon (Mann-Whitney)

8. Primary Outcome: Caregiver Affect Measured by the Joint Engagement Rating Inventory (JERI)
Description: as for outcome 6
Time Frame: Baseline and Follow-up (after 12 intervention sessions, up to 3 months)
Population: as for outcome 1
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Caregiver-Child Dyads With ASD (In-person Intervention ONLY) | Caregiver-Child Dyads With ASD (Telehealth Intervention) | Children With Typical Development | Children With Developmental Delay
Number analyzed (Participants) | 8 | 9 | 2 | 1
score on a scale
  Baseline | 4 [4 to 5] | 5 [4 to 7] | 5 [5 to 5] | 3 [3 to 3]
  Follow-up: number analyzed (Participants) | 8 | 9 | 0 | 0
  Follow-up | 4.5 [4 to 6] | 5 [4 to 7] |  |

9. Primary Outcome: Initiation of Joint Attention (IJA) Measured by the Early Social Communication Scales (ESCS)
Description: Joint attention skills will be measured using the Early Social Communication Scales (ESCS) in the ASD group; the typically developing group; and the developmental delay group. The ESCS assesses nonverbal communication skills, is normed for typically developing children 18 to 30 months of age in addition to children with developmental delay expressive language level is in approximately the same range. Frequency scores for initiation of joint attention (IJA) will be derived from behavioral observations during a series of tasks presented by an examiner blind to child diagnosis. IJA score ranges from 0 to 100 where a higher value indicates greater initiation of joint attention.
Time Frame: Baseline
Population: Only applicable to Caregiver-Child Dyads With ASD, Children with typical development, and Children with developmental delay groups. This measure was introduced later in the study and therefore not administered to all participants. Data not collected on the Caregiver-Child Dyads With ASD (Telehealth Intervention) group.
Measure: Mean (Full Range); unit: score on a scale
Groups:
- Caregiver-Child Dyads With ASD (In-person Intervention): Participants in this arm will be caregivers of and children with ASD. Early Start Denver Model (ESDM): Twelve one hour sessions, skill is introduced by "Help is in your hands" Community ESDM videos. Session skills include specific strategies caregivers can use to increase their child's attention to people and their child's communication; strategies to identify, create and use joint activity routines to engage with and teach their child; in addition to ways to use the ABCs of learning to teach their child new behaviors. "Help is in your hands" Community ESDM materials also provide video examples of other caregivers using the session skill with their child. The early childhood development practitioner then coaches the caregiver in the session skill, in at least two activities. The goal of coaching was to provide enough support for the caregiver to experience success in implementing the new skill with their child. Coaching is followed by caregiver reflection and a discussion of generalization of the new skill across various daily activities, using a daily activities visual aid.
- Caregiver-Child Dyads With ASD (Telehealth Intervention): Participants in this arm will be caregivers of and children with ASD receiving telehealth intervention (adaptation due to COVID-19 restrictions).
  Telehealth coaching: The telehealth coaching intervention was informed by the Community-Early Start Denver Model (C-ESDM) materials. Twelve session-specific visuals with simple-text (for caregivers) and session scripts (for non-specialist coaches) were developed by the research team. Over 12, 1-hour asynchronous caregiver coaching sessions that are delivered by non-specialists, caregivers were coached in strategies to increase child attention to their social world, increase child communication, create and build joint activity routines, and understand and use the ABCs to support the development of new behaviors. The session itself being delivered via phone. Prior to the coaching session staff shared session materials with the family via WhatsApp. Prior to the session the caregiver shared a 6-min video of an interaction with their child. During the session, the caregiver and coach reviewed the video, and the caregiver completed a self-reflection checklist.
Arm/Group | Caregiver-Child Dyads With ASD (In-person Intervention) | Caregiver-Child Dyads With ASD (Telehealth Intervention) | Children With Typical Development | Children With Developmental Delay
Number analyzed (Participants) | 9 | 0 | 1 | 1
score on a scale | 8.33 [0 to 19] |  | 69 [69 to 69] | 27 [27 to 27]

10. Primary Outcome: Response to Joint Attention (RJA) Measured by the Early Social Communication Scales (ESCS)
Description: Joint attention skills will be measured using the Early Social Communication Scales (ESCS) in the ASD group; the typically developing group; and the developmental delay group. The ESCS assesses nonverbal communication skills, is normed for typically developing children 18 to 30 months of age in addition to children with developmental delay expressive language level is in approximately the same range. Frequency scores for response to joint attention (RJA) will be derived from behavioral observations during a series of tasks presented by an examiner blind to child diagnosis. RJA score ranges from 0 to 20 where a higher value indicates greater response to joint attention.
Time Frame: Baseline
Population: as for outcome 9
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Caregiver-Child Dyads With ASD (In-person Intervention) | Caregiver-Child Dyads With ASD (Telehealth Intervention) | Children With Typical Development | Children With Developmental Delay
Number analyzed (Participants) | 9 | 0 | 1 | 1
score on a scale | 5 [1 to 13] |  | 15 [15 to 15] | 7 [7 to 7]

11. Primary Outcome: Language and Communication Developmental Quotient on the Griffiths Scales of Child Development 3rd Edition (Griffiths-III)
Description: The Griffiths Scales of Child Development, Third Edition (Griffiths III) is a comprehensive, developmental measure for continuous use from birth to 5 years 11 months (71 months). Although not standardized in South Africa (standardization samples are from the United Kingdom and Ireland), this developmental assessment is widely used in South Africa. The Griffiths III provides an overall measure of a child's development, as well as an individual profile of strengths and needs across five areas: Foundations of Learning; Language and Communication; Eye and Hand Coordination; Personal-Social-Emotional; and Gross Motor. Developmental quotients (DQs) were calculated by (Developmental Age/Chronological Age) *100. Griffiths III DQs range from 1 to 100 where higher scores indicate that the child performs at or near expected chronological age as compared with a normative sample of children the same age.
Time Frame: Baseline and Follow up (after 12 intervention sessions, up to 3 months)
Population: Participants who completed the study. Only applicable to child groups. Data not collected on Caregiver-Child Dyads With ASD (Telehealth Intervention) - Children group. Data only collected at baseline for Children with Typical Development and Children with Developmental Delay.
Measure: Median (Full Range); unit: units on a scale
Groups:
- Caregiver-Child Dyads With ASD (Telehealth Intervention) - Children: Participants in this arm will be children with ASD receiving telehealth intervention (adaptation due to COVID-19 restrictions) or as a continuation of in-person intervention.
  Telehealth coaching: The telehealth coaching intervention was informed by the Community-Early Start Denver Model (C-ESDM) materials. Twelve session-specific visuals with simple-text (for caregivers) and session scripts (for non-specialist coaches) were developed by the research team. Over 12, 1-hour asynchronous caregiver coaching sessions that are delivered by non-specialists, caregivers were coached in strategies to increase child attention to their social world, increase child communication, create and build joint activity routines, and understand and use the ABCs to support the development of new behaviors. The session itself being delivered via phone. Prior to the coaching session staff shared session materials with the family via WhatsApp. Prior to the session the caregiver shared a 6-min video of an interaction with their child. During the session, the caregiver and coach reviewed the video, and the caregiver completed a self-reflection checklist.
Arm/Group | Caregiver-Child Dyads With ASD (In-person Intervention ONLY) - Children | Caregiver-Child Dyads With ASD (Telehealth Intervention) - Children | Children With Typical Development | Children With Developmental Delay
Number analyzed (Participants) | 8 | 0 | 2 | 1
units on a scale
  Baseline | 57.73 [51.16 to 64.06] |  | 114 [NA to NA] — Unable to calculate IQR due to insufficient number of participants/values. | 50 [NA to NA] — Unable to calculate IQR due to insufficient number of participants/values.
  Follow-up: number analyzed (Participants) | 8 | 0 | 0 | 0
  Follow-up | 62.24 [51.28 to 70.69] |  |  |
Statistical Analysis 1: Comparison: Caregiver-Child Dyads With ASD (In-person Intervention ONLY) - Children; Test type: Other; p = 0.004, Wilcoxon (Mann-Whitney)

12. Primary Outcome: Personal-Social-Emotional Developmental Quotient on the Griffiths Scales of Child Development 3rd Edition (Griffiths-III)
Description: as for outcome 11
Time Frame: Baseline and Follow up (after 12 intervention sessions, up to 3 months)
Population: as for outcome 11
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Caregiver-Child Dyads With ASD (In-person Intervention ONLY) - Children | Caregiver-Child Dyads With ASD (Telehealth Intervention) - Children | Children With Typical Development | Children With Developmental Delay
Number analyzed (Participants) | 8 | 0 | 2 | 1
units on a scale
  Baseline | 63.41 [53.49 to 71.43] |  | 115 [NA to NA] — Unable to calculate IQR due to insufficient number of participants/values. | 83.33 [NA to NA] — Unable to calculate IQR due to insufficient number of participants/values.
  Follow-up: number analyzed (Participants) | 8 | 0 | 0 | 0
  Follow-up | 65.53 [58.33 to 73.91] |  |  |
Statistical Analysis 1: Comparison: Caregiver-Child Dyads With ASD (In-person Intervention ONLY) - Children; Test type: Other; p = 0.084, Wilcoxon (Mann-Whitney)

13. Primary Outcome: Socialization Subscale Standard Score on the Vineland Adaptive Behavior Scales - 3rd Edition (VABS-3)
Description: The Vineland Adaptive Behavior Scales, Third Edition (Vineland-3) is an individually-administered measure of adaptive behavior that is widely used to assess individuals with intellectual, developmental, and other disabilities. The Vineland-3 contains 5 domains each with 2-3 subdomains. The main domains are: Communication, Daily Living Skills, Socialization, Motor Skills, and Maladaptive Behavior. The Caregiver Interview Form uses the Vineland semistructured interview technique to elicit information about the examinee's adaptive functioning from a parent or caregiver. Item responses are collected on a 3-point Likert scale with values representing 0 (never), 1 (sometimes), and 2 (usually or often) to capture frequency of target behavior. Some items require binary responses (yes/no). The VABS-3 Socialization subscale score ranges from 20-140 where a higher score indicates greater frequency of target behavior.
Time Frame: Baseline and Follow up (after 12 intervention sessions, up to 3 months)
Population: Participants who completed the study. Only applicable to the Caregiver-Child Dyads With ASD groups.
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Caregiver-Child Dyads With ASD (In-person Intervention ONLY) | Caregiver-Child Dyads With ASD (Telehealth Intervention)
Number analyzed (Participants) | 8 | 9
score on a scale
  Baseline | 61 [42 to 77] | 63 [46 to 73]
  Follow-up | 67.5 [42 to 84] | 61 [54 to 73]
Statistical Analysis 1: Comparison: Caregiver-Child Dyads With ASD (In-person Intervention ONLY); Test type: Other; p = 0.42, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Caregiver-Child Dyads With ASD (Telehealth Intervention); Test type: Other; p = 0.171, Wilcoxon (Mann-Whitney)

14. Primary Outcome: Communication Subscale Standard Score on the Vineland Adaptive Behavior Scales - 3rd Edition (VABS-3)
Description: The Vineland Adaptive Behavior Scales, Third Edition (Vineland-3) is an individually-administered measure of adaptive behavior that is widely used to assess individuals with intellectual, developmental, and other disabilities. The Vineland-3 contains 5 domains each with 2-3 subdomains. The main domains are: Communication, Daily Living Skills, Socialization, Motor Skills, and Maladaptive Behavior. The Caregiver Interview Form uses the Vineland semistructured interview technique to elicit information about the examinee's adaptive functioning from a parent or caregiver. Item responses are collected on a 3-point Likert scale with values representing 0 (never), 1 (sometimes), and 2 (usually or often) to capture frequency of target behavior. Some items require binary responses (yes/no). The VABS-3 Communication subscale score ranges from 20-140 where a higher score indicates greater frequency of target behavior.
Time Frame: Baseline and Follow up (after 12 intervention sessions, up to 3 months)
Population: Participants who completed the study. Only applicable to the Caregiver-Child Dyads With ASD groups.
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Caregiver-Child Dyads With ASD (In-person Intervention ONLY) | Caregiver-Child Dyads With ASD (Telehealth Intervention)
Number analyzed (Participants) | 8 | 9
score on a scale
  Baseline | 41 [26 to 62] | 34 [20 to 76]
  Follow-up | 50 [28 to 64] | 40 [32 to 70]
Statistical Analysis 1: Comparison: Caregiver-Child Dyads With ASD (In-person Intervention ONLY); Test type: Other; p = 0.011, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Caregiver-Child Dyads With ASD (Telehealth Intervention); Test type: Other; p = 0.049, Wilcoxon (Mann-Whitney)

15. Secondary Outcome: Acceptability of Telehealth Intervention (as Measured by the Acceptability of Intervention Measure, AIM)
Description: A 5-item scale that measures the extent to which a new treatment, or an innovation, can be successfully used or carried out within a given agency or setting. Scores are indicated on a scale of 1 - 5 with higher scores indicating greater acceptability.
Time Frame: Follow-up (within 2 weeks of ending sessions)
Population: Participants who completed the study. Only applicable to Caregiver-Child Dyads With ASD (Telehealth Intervention) - Caregivers, Early Childhood Development (ECD) Practitioners and ECD Practitioner School Supervisors, and Early Start Denver Model (ESDM) Supervisors groups.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Caregiver-Child Dyads With ASD (Telehealth Intervention) - Caregivers: Participants in this arm will be caregivers of children with ASD receiving telehealth intervention (adaptation due to COVID-19 restrictions) or as a continuation of in-person intervention.
  Telehealth coaching: The telehealth coaching intervention was informed by the Community-Early Start Denver Model (C-ESDM) materials. Twelve session-specific visuals with simple-text (for caregivers) and session scripts (for non-specialist coaches) were developed by the research team. Over 12, 1-hour asynchronous caregiver coaching sessions that are delivered by non-specialists, caregivers were coached in strategies to increase child attention to their social world, increase child communication, create and build joint activity routines, and understand and use the ABCs to support the development of new behaviors. The session itself being delivered via phone. Prior to the coaching session staff shared session materials with the family via WhatsApp. Prior to the session the caregiver shared a 6-min video of an interaction with their child. During the session, the caregiver and coach reviewed the video, and the caregiver completed a self-reflection checklist.
Arm/Group | Caregiver-Child Dyads With ASD (Telehealth Intervention) - Caregivers | Early Childhood Development (ECD) Practitioners and ECD Practitioner School Supervisors | Early Start Denver Model (ESDM) Supervisors
Number analyzed (Participants) | 9 | 3 | 3
score on a scale | 4.25 (0.4) | 4.66 (0.6) | 4.78 (0.1)

16. Secondary Outcome: Appropriateness of Telehealth Intervention (as Measured by the Intervention Appropriateness Measure, IAM)
Description: A 5-item scale that measures the extent to which a new treatment, or an innovation, can be successfully used or carried out within a given agency or setting. Scores are indicated on a scale of 1-5 with higher scores indicating greater appropriateness.
Time Frame: Follow-up (within 2 weeks of ending sessions)
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Caregiver-Child Dyads With ASD (Telehealth Intervention) - Caregivers | Early Childhood Development (ECD) Practitioners and ECD Practitioner School Supervisors | Early Start Denver Model (ESDM) Supervisors
Number analyzed (Participants) | 9 | 3 | 3
score on a scale | 4.47 (0.4) | 4.66 (0.6) | 4.66 (0.8)

17. Secondary Outcome: Feasibility of Intervention (as Measured by the Feasibility of Intervention Measure, FIM)
Description: A 5-item scale that measures the extent to which a new treatment, or an innovation, can be successfully used or carried out within a given agency or setting. Scores are indicated on a scale of 1-5 with higher scores indicating greater feasibility.
Time Frame: Follow-up (within 2 weeks of ending sessions)
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Caregiver-Child Dyads With ASD (Telehealth Intervention) - Caregivers | Early Childhood Development (ECD) Practitioners and ECD Practitioner School Supervisors | Early Start Denver Model (ESDM) Supervisors
Number analyzed (Participants) | 9 | 3 | 3
score on a scale | 4.14 (0.4) | 4.66 (0.6) | 4.9 (0.1)

18. Secondary Outcome: Fidelity of Intervention Delivery, as Measured by the Caregiver ESDM Fidelity Rating System
Description: ESDM Fidelity Rating System uses a 13 item rating scale that includes ratings of performance on core intervention strategies from 1 to 5 (1 represents a lack of an effective display of the practices specified, and 5 represents the best possible example of this teaching behavior). Fidelity of implementation of Naturalistic Developmental Behavioral Intervention (NDBI) strategies will be manually coded by certified ESDM therapists. Mean fidelity scores (with SD) will be calculated across study participants in order to assess change in NDBI strategies. ESDM Fidelity Rating System scores range from 0 to 100 with a higher score reflecting interactions closer to ESDM principles.
Time Frame: Baseline and Follow-up (up to 4 months)
Population: Participants who completed the study. Only applicable to the Caregiver-Child Dyads With ASD Caregiver groups.
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Caregiver-Child Dyads With ASD (In-person Intervention ONLY) - Caregivers | Caregiver-Child Dyads With ASD (Telehealth Intervention) - Caregivers
Number analyzed (Participants) | 8 | 9
score on a scale
  Baseline | 60 [45 to 67] | 55 [44 to 78]
  Follow-up | 75 [65 to 87] | 68 [53 to 83]
Statistical Analysis 1: Comparison: Caregiver-Child Dyads With ASD (In-person Intervention ONLY) - Caregivers; Test type: Other; p = 0.003, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Caregiver-Child Dyads With ASD (Telehealth Intervention) - Caregivers; Test type: Other; p = 0.139, Wilcoxon (Mann-Whitney)

19. Other Pre Specified Outcome: Postural Sway Measured by the SenseToKnow App
Description: SenseToKnow is an app developed for mobile devices that is designed to elicit autism risk behaviors. In order to administer the app, children sit on the parent's lap with the mobile device at eye level for the child. The app is comprised of a set of stimuli (videos and games) that are designed to elicit autism spectrum disorder (ASD) symptoms, such as facial expressions. Multi-modal time-series video-frame-level data streams from the computer vision analysis output of SenseToKnow will be summarized with descriptive statistics and visualizations. We extract landmarks and determine the correct features from them to yield precise measurements of attention, gaze, affect, and posture. Each computer vision analysis feature will be transformed into one or more binary, count, or continuous participant-level summary variable (for e.g. number of times orienting to name).
Time Frame: Baseline and Baseline and Follow up (after 12 intervention sessions, up to 3 months) ASD group; Baseline typically developing and developmental delay group
Reporting Status: Not Posted

20. Other Pre Specified Outcome: Gaze Patterns Measured by the SenseToKnow App
Description: as for outcome 19
Time Frame: as for outcome 19
Reporting Status: Not Posted

21. Other Pre Specified Outcome: Social Referencing Measured by the SenseToKnow App
Description: as for outcome 19
Time Frame: as for outcome 19
Reporting Status: Not Posted

22. Other Pre Specified Outcome: Affective Response Measured by the SenseToKnow App
Description: as for outcome 19
Time Frame: Baseline and fBaseline and Follow up (after 12 intervention sessions, up to 3 months) ASD group; Baseline typically developing and developmental delay group
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Up to 4 months
Arm/Group | Caregiver-Child Dyads With ASD (In-person Intervention ONLY) - Caregivers | Caregiver-Child Dyads With ASD (In-person Intervention ONLY) - Children | Caregiver-Child Dyads With ASD (In-person, Then Telehealth Intervention) - Caregivers | Caregiver-Child Dyads With ASD (In-person, Then Telehealth Intervention) - Children | Caregiver-Child Dyads With ASD (Telehealth Intervention ONLY) - Caregivers | Caregiver-Child Dyads With ASD (Telehealth Intervention ONLY) - Children | Children With Typical Development | Children With Developmental Delay | Early Childhood Development (ECD) Practitioners and ECD Practitioner School Supervisors | Early Start Denver Model (ESDM) Supervisors
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/17 | 0/2 | 0/2 | 0/12 | 0/12 | 0/2 | 0/1 | 0/4 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/17 | 0/2 | 0/2 | 0/12 | 0/12 | 0/2 | 0/1 | 0/4 | 0/3
Other Adverse Events (participants affected / at risk) | 0/17 | 0/17 | 0/2 | 0/2 | 0/12 | 0/12 | 0/2 | 0/1 | 0/4 | 0/3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-07-26): https://cdn.clinicaltrials.gov/large-docs/88/NCT04068688/Prot_SAP_001.pdf
  • Informed Consent Form (2021-07-09): https://cdn.clinicaltrials.gov/large-docs/88/NCT04068688/ICF_000.pdf